CLINICAL TRIAL: NCT05332262
Title: Ability of a Precision Medicine Approach to Identify Stable CAD Patients Undergoing Elective PCI Who Are at Risk of Peri-PCI Myocardial Infarction/Myocardial Injury: The ABCD-Gene Prospective Study
Brief Title: A Precision Medicine Approach to Identify Patients Undergoing Elective PCI at Risk of Peri-PCI Myocardial Infarction
Status: Recruiting | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB202200298
Record Dates: First submitted 2022-04-11; First posted 2022-04-18 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease
Keywords: percutaneous coronary intervention; clopidogrel; high platelet reactivity; myocardial injury
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be stored for future analysis, which may include assessment of markers of inflammation, novel genetic variants, or micro-RNA. Blood samples will be stored in a UF-approved storage bank (IRB202100157).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High ABCD-GENE score (≥10): All patients in this cohort will have an ABCD-GENE score ≥10 and will be receiving clopidogrel following PCI as per standard of care.
  The ABCD-GENE score encompasses a total of 5 variables: 4 clinical (age, body mass index, chronic kidney disease status, and diabetes mellitus) and 1 genetic (CYP2C19 LOF).
  Interventions: Diagnostic Test: Assessment of platelet reactivity; Diagnostic Test: Troponin measurement
- Low ABCD-GENE score (<10): All patients in this cohort will have an ABCD-GENE score <10 and will be receiving clopidogrel following PCI as per standard of care.
  The ABCD-GENE score encompasses a total of 5 variables: 4 clinical (age, body mass index, chronic kidney disease status, and diabetes mellitus) and 1 genetic (CYP2C19 LOF).
  Interventions: Diagnostic Test: Assessment of platelet reactivity; Diagnostic Test: Troponin measurement

INTERVENTIONS:
Diagnostic Test: Assessment of platelet reactivity — Assessment of platelet reactivity and HPR status will be performed post-PCI. Platelet reactivity will be measured by VerifyNow P2Y12 and HPR status will be defined using a cut-off value of platelet reactivity units (PRU)>208.
Diagnostic Test: Troponin measurement — Measurement of high sensitivity troponin for the assessment for the presence of myocardial infarction/myocardial injury will be performed post-PCI.

SUMMARY:
Despite the relative safety of PCI with new generation stents, peri-PCI thrombotic complications, including myocardial infarction and myocardial injury, are common in elective PCI, occurring in up to 30% of patients. Importantly, these events are associated with poor prognosis. The risk of peri-PCI myocardial infarction/myocardial injury has been in part attributed to HPR. The aim of this study is to prospectively validate the accuracy of the ABCD-GENE score in identifying stable CAD patients undergoing elective PCI treated with standard of care clopidogrel who are at risk of peri-PCI myocardial infarction/myocardial injury. This investigation will be a prospective cohort study conducted in a population of patients (n=500) with stable CAD undergoing elective PCI treated with standard of care clopidogrel. By integrating genetic data with clinical variables, patients will be stratified into 2 cohorts based on their ABCD-GENE score (using a cut-off of 10). Assessments to define HPR status and myocardial infarction/myocardial injury will be performed post-PCI.

DETAILED DESCRIPTION:
Antiplatelet therapy with aspirin and a P2Y12 inhibitor is the cornerstone of treatment for patients undergoing percutaneous coronary intervention (PCI). Clopidogrel is the recommended P2Y12 inhibitor in patients with stable coronary artery disease (CAD) undergoing elective PCI. However, clopidogrel effects are subject to variability and 30-40% of patients have high platelet reactivity (HPR), which translates into higher rates of thrombotic complications. Despite the relative safety of PCI with new generation stents, peri-PCI thrombotic complications, including myocardial infarction and myocardial injury, are common in elective PCI, occurring in up to 30% of patients. Importantly, these events are associated with poor prognosis. The risk of peri-PCI myocardial infarction/myocardial injury has been in part attributed to HPR. The investigators recently developed a precision medicine tool integrating clinical and genetic factors called ABCD-GENE able to identify HPR status. This score helps characterize patients at risk for peri-PCI thrombotic complications, who can thus potentially benefit from changes in antiplatelet treatment regimen. However, the ABCD-GENE score was generated through retrospective assessments, thus warranting prospective validation. The high frequency of elective PCI procedures and the prevalence with which myocardial infarction/myocardial injury occurs underscore the need for tools that can better identify patients at risk so that therapeutic measures can be implemented to improve their prognosis. The aim of this study is to prospectively validate the accuracy of the ABCD-GENE score in identifying stable CAD patients undergoing elective PCI treated with standard of care clopidogrel who are at risk of peri-PCI myocardial infarction/myocardial injury. This investigation will be a prospective cohort study conducted in a population of patients (n=500) with stable CAD undergoing elective PCI treated with standard of care clopidogrel. By integrating genetic data with clinical variables, patients will be stratified into 2 cohorts based on their ABCD-GENE score (using a cut-off of 10). Assessments to define HPR status and myocardial infarction/myocardial injury will be performed post-PCI.

ELIGIBILITY:
Inclusion criteria:

1. Stable CAD undergoing elective PCI;
2. Male or females, Age ≥ 18 years old;
3. Troponin negative before PCI*;
4. Background of aspirin therapy;

   * If troponin is unknown before coronary angiography and no clinical signs of acute coronary syndrome is present, a troponin will not be collected as this is line with standard practice.

Exclusion criteria:

1. Current presentation with myocardial infarction;
2. On treatment with prasugrel or ticagrelor;
3. Documented hypersensitivity to clopidogrel;
4. Use of an intravenous antiplatelet therapy (i.e., cangrelor or GPI) during PCI;
5. Unable to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All-comers population of troponin-negative CAD patients undergoing elective PCI as part of their standard of care at the Division of Cardiology of University of Florida Health, Jacksonville, Florida. Genotyping will be performed as per standard of care in the UF Health Pathology lab.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Peri-PCI myocardial infarction or myocardial injury | 24 hours
  The primary endpoint of the study will be rate of peri-PCI myocardial infarction or myocardial injury, which will be compared between the high ABCD-GENE score cohort and the low ABCD-GENE score cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Franchi, MD, Principal Investigator — University of Florida College of Medicine Jacksonville
Locations (1):
- University of Florida Jacksonville, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No